CLINICAL TRIAL: NCT01780844
Title: A Phase 2a, Randomized, Open-label, Active Control, Multi-Center Study to Assess the Efficacy and Safety of ASKP1240 in de Novo Kidney Transplant Recipients
Brief Title: A Study to Assess the Efficacy and Safety of ASKP1240 in de Novo Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7163-CL-0108
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; de novo Kidney Transplantation; ASKP1240
MeSH Terms: interventions — bleselumab; Tacrolimus; Mycophenolic Acid; Basiliximab; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Active Comparator): Basiliximab induction + Tacrolimus + MMF + Corticosteroids
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil (MMF); Drug: Basiliximab; Drug: Methylprednisone; Drug: Prednisone
- CNI avoidance (Experimental): Basiliximab induction + ASKP1240 + MMF + Corticosteroids
  Interventions: Drug: ASKP1240; Drug: Mycophenolate Mofetil (MMF); Drug: Basiliximab; Drug: Methylprednisone; Drug: Prednisone
- CNI minimization-MMF avoidance (Experimental): Basiliximab induction + ASKP1240 + Tacrolimus + Corticosteroids
  Interventions: Drug: ASKP1240; Drug: Tacrolimus; Drug: Basiliximab; Drug: Methylprednisone; Drug: Prednisone

INTERVENTIONS:
Drug: ASKP1240 — intravenous infusion
  Arms: CNI avoidance; CNI minimization-MMF avoidance
Drug: Tacrolimus — intravenous or oral
  Other Names: Prograf®
  Arms: CNI minimization-MMF avoidance; Standard of Care
Drug: Mycophenolate Mofetil (MMF) — intravenous or oral
  Other Names: CellCept®
  Arms: CNI avoidance; Standard of Care
Drug: Basiliximab — intravenous
  Other Names: Simulect®
Drug: Methylprednisone — Intravenous
Drug: Prednisone — Oral

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ASKP1240, an anti-CD40 monoclonal antibody, for the prophylaxis of organ rejection after kidney transplantation. This study will compare the efficacy of basiliximab induction, ASKP1240, mycophenolate mofetil (MMF), and steroids [calcineurin inhibitor (CNI) avoidance] to the standard of care immunosuppressive regimen (basiliximab induction + tacrolimus + MMF + steroids). In addition, the study will compare the efficacy of basiliximab induction, ASKP1240, tacrolimus and steroids [CNI minimization-MMF avoidance] to the standard of care immunosuppressive regimen (basiliximab induction + tacrolimus + MMF + steroids).

DETAILED DESCRIPTION:
Subjects will be followed for 6 months. Upon completion of the first 6 months of the study, subjects may participate in the Long Term Extension period of the study. Subjects will remain on their original treatment arm up to three years post-transplant (and / or Sponsor discontinues development or the subject no longer wishes to participate in the study).

ELIGIBILITY:
Inclusion Criteria:

* Subject is a recipient of a de novo kidney from a living or deceased donor

Exclusion Criteria:

* Subject has induction therapy, other than study-assigned basiliximab, planned as part of initial immunosuppressive regimen
* Subject has previously received or is receiving an organ transplant other than a kidney
* Subject will receive a solitary kidney from a deceased donor < 5 years of age
* Subject will receive a kidney with an anticipated cold ischemia time (CIT) of > 30 hours
* Subject will receive a kidney that meets both Extended Criteria Donor (ECD) and Donation after Cardiac Death (DCD) criteria. Note: a kidney that meets either ECD or DCD criteria is eligible for inclusion
* Subject will receive an ABO incompatible donor kidney
* Subject has a current calculated panel reactive antibody (cPRA) level >50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2013-03-05 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
Biopsy-proven acute (T or B cell) rejection (BPAR) (Banff 2007 Grade ≥ 1) by local review | 6 months

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) | 6 months
  GFR is based on Modification of Diet in Renal Disease (4 variable-MDRD) criteria
Patient Survival | 6 months
  Subject survival is defined as any subject who does not die during the study.
Graft Survival | 6 months
  Graft survival is defined as any subject who does not experience graft loss during the study. Graft loss is defined as subject death, retransplantation, transplant nephrectomy, or the permanent return to dialysis (greater than 30 days).

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (42):
- United States (42):
  - Site US10006, Birmingham, Alabama
  - Site US10024, Phoenix, Arizona
  - Site US10008, Los Angeles, California
  - Site US10021, Palo Alto, California
  - Site US10030, San Diego, California
  - Site US10004, San Francisco, California
  - Site US10003, San Francisco, California
  - Site US10013, Aurora, Colorado
  - Site US10007, Atlanta, Georgia
  - Site US10041, Augusta, Georgia
  - Site US10010, Chicago, Illinois
  - Site US10018, Chicago, Illinois
  - Site US10037, Chicago, Illinois
  - Site US10015, Lexington, Kentucky
  - Site US10045, New Orleans, Louisiana
  - Site US10014, Baltimore, Maryland
  - Site US10017, Ann Arbor, Michigan
  - Site US10025, St Louis, Missouri
  - Site US10022, Livingston, New Jersey
  - Site US10031, Buffalo, New York
  - Site US10034, New York, New York
  - Site US10023, New York, New York
  - Site US10019, The Bronx, New York
  - Site US10036, Chapel Hill, North Carolina
  - Site US10042, Charlotte, North Carolina
  - Site US10016, Durham, North Carolina
  - Site US10026, Greenville, North Carolina
  - Site US10009, Cincinnati, Ohio
  - Site US10040, Cleveland, Ohio
  - Site US10032, Cleveland, Ohio
  - Site US10027, Harrisburg, Pennsylvania
  - Site US10038, Pittsburgh, Pennsylvania
  - Site US10012, Charleston, South Carolina
  - Site US10028, Memphis, Tennessee
  - Site US10035, Nashville, Tennessee
  - Site US10001, Dallas, Texas
  - Site US10002, Fort Worth, Texas
  - Site US10029, Houston, Texas
  - Site US10044, Houston, Texas
  - Site US10033, Salt Lake City, Utah
  - Site US10020, Charlottesville, Virginia
  - Site US10005, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency.

REFERENCES:
- [Derived] Harland RC, Klintmalm G, Jensik S, Yang H, Bromberg J, Holman J, Kumar MSA, Santos V, Larson TJ, Wang X. Efficacy and safety of bleselumab in kidney transplant recipients: A phase 2, randomized, open-label, noninferiority study. Am J Transplant. 2020 Jan;20(1):159-171. doi: 10.1111/ajt.15591. Epub 2019 Oct 19. PMID 31509331
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/7163-CL-0108/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=25564&tenant=MT_AST_9011